CLINICAL TRIAL: NCT02882126
Title: An Open-Label Extension Trial to Evaluate the Safety of Continued Therapy With Subcutaneous Remodulin® in Subjects With Pulmonary Arterial Hypertension Who Completed Study CVT-CV-003
Brief Title: An Open Label Extension Study to Evaluate the Safety of Continued Therapy of Subcutanous Remodulin® in Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision
Sponsor: United Therapeutics (Industry)
Collaborators: CVie Therapeutics Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVT-CV-004
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Subcutaneous Treprostinil; Remodulin; 6 Minute Walk Test
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subcutaneous Treprostinil (Experimental): Open-label access; The initial dose of Remodulin for this study will be the same as each subject's final dose in study CVT-CV-003. Dose modification will be based according to clinical response and tolerability.
  Interventions: Drug: Subcutaneous Treprostinil

INTERVENTIONS:
Drug: Subcutaneous Treprostinil — Remodulin (1.0, 2.5, 5 and 10 mg/ml formulations as available) will be administered by continuous subcutaneous infusion via a subcutaneous cannula using a microbore infusion tubing set and a micro infusion pump.
  Other Names: Remodulin

SUMMARY:
This is a multicenter, open-label trial to evaluate the safety of continued therapy with subcutaneous Remodulin® in subjects with pulmonary arterial hypertension (PAH) who complete the CVT-CV-003 study. The study will include about 50 subjects at up to 10 clinical trial centers in China who completed all required assessments in the CVT-CV-003 study. Study visits for data collection will occur at month 6 and 12 with yearly visits beyond 12 months until the study is discontinued by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible for inclusion in this study if all of the following criteria apply:

1. The subject voluntarily gives written informed consent to participate in the study.
2. The subject participated in and completed study CVT-CV-003.
3. Sexually active women of childbearing potential must practice true abstinence from intercourse when it is in line with their preferred and usual lifestyle, or use two different forms of highly effective contraception. Medically acceptable forms of effective contraception include: (1) approved hormonal contraceptive (such as birth control pills), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, (3) an intrauterine device (IUD), or (4) partner vasectomy. Women of child bearing potential include any females who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or are not postmenopausal (defined as amenorrhea for at least 12 consecutive months).

   Males participating in the study must use a condom during the length of the study, and for at least 48 hours after discontinuing study medication.
4. The subject has not developed a concurrent illness or condition during the conduct of the previous study (including but not restricted to, sleep apnea, chronic renal insufficiency, anemia, uncontrolled systemic hypertension or left sided heart disease) that would make participation in this study detrimental to the subject's health in the opinion of the Investigator.
5. In the opinion of the Principal Investigator, the subject is able to communicate effectively with study personnel, is considered reliable, willing and likely to be cooperative with protocol requirements, including attending all study visits, and is mentally and physically capable of administering Remodulin by continuous SC infusion using a micro infusion pump.

Exclusion Criteria:

A subject is not eligible for inclusion in this study if any of the following criteria apply:

1. The subject permanently discontinued Remodulin during study CVT-CV-003.
2. The subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Among Subjects through Study Completion | Study Completion, an Average of 3 Years
  Adverse events among participants will be recorded throughout participation in the study. The incidence of adverse events among subjects through study completion, an average of 3 years, will be described by the number of subjects analyzed and the percentage of those subjects who experienced an adverse event until study completion.
Change in 6-minute Walk Distance (6MWD) From Baseline to Month 12 | Baseline and Month 12
  The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out activities of daily living. Change in 6MWD from Baseline to Month 12, correlates with the current clinical standard for assessing patient functional status in the treatment of PAH and is considered an objective measure of patient functional status. Subjects will be instructed to walk down a corridor at a comfortable speed as far as they can manage for six minutes. Distance <500 meters suggests considerable exercise limitation; Distance 500-800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation.
Change in Borg Dyspnea Score (following 6MWT) from Baseline to Month 12 | Baseline and Month 12
  The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea (difficulty in breathing) experienced during the six-minute walk test (6MWT). The Borg dyspnea score will be assessed immediately following the 6MWT. Scores range from 0 (for no shortness of breath) to 10 (for the greatest shortness of breath ever experienced). Changes from Baseline to Month 12 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.
Number of Participants with a Change from Baseline World Health Organization (WHO) Functional Classification at Month 12 | Change from Baseline at Month 12
  The WHO Functional Class of pulmonary hypertension is a physical activity rating scale as follows: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms. Changes from Baseline to Month 12 will be summarized and compared between treatment groups using descriptive statistics. No formal hypothesis testing will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Zhongshan Hospital affiliated with Fudan University
Locations (10):
- China (10):
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Fu Wai Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Xiangya Hospital Centre South University, Changsha
  - Guangdong General Hospital, Guangzhou
  - Zhongshan Hospital affiliated with Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Wuhan Asia Heart Hospital, Wuhan